CLINICAL TRIAL: NCT07015853
Title: IIT2024-02-SHIAO-ASTRAEA: ReinvigorAting ReSponse To ImmunotheRApy in MEtAstatic TNBC With Combination Myeloid Inhibition and Radiation
Brief Title: ASTRAEA: ReinvigorAting ReSponse To ImmunotheRApy in MEtAstatic TNBC With Combination Myeloid Inhibition and Radiation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Shiao (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Stephen Shiao, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024-02-SHIAO-ASTRAEA
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: TNBC - Triple-Negative Breast Cancer; Breast Cancer
Keywords: Pembrolizumab; Axatilimab; CSF-1R inhibitor; potent humanized immunoglobulin G4 (IgG4); Radiation Therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — pembrolizumab; Radiotherapy; axatilimab

STUDY DESIGN:
Intervention Model Description: Open label, single-arm, prospective therapeautic trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab, Radiotherapy, Axatilimab (Experimental): Pembrolizumab (MK-3475), 200 mg IV Q3W starting at C1D1/Week 1 for up to 2 years, until disease progression, or treatment intolerance.
  Radiotherapy, 8 Gy x 3 fractions over 3 consecutive days at C1D8/Week 2; Axatilimab (SNDX-6352; INCA034176), 1 mg/kg, IV, Q2W starting 1 week post- RT C1D15/Week 3 until disease progression or treatment intolerance.
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy; Drug: Axatilimab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (MK-3475), 200 mg IV Q3W starting at C1D1/Week 1 for up to 2 years, until disease progression, or treatment intolerance.
  Other Names: Ketruda
Radiation: Radiotherapy — RT, 8 Gy x 3 fractions over 3 consecutive days at C1D8/Week 2;
Drug: Axatilimab — Axatilimab (SNDX-6352; INCA034176), 1 mg/kg, IV, Q2W starting 1 week post- RT C1D15/Week 3 until disease progression or treatment intolerance.
  Other Names: CSF-1R inhibitor

SUMMARY:
Open label, single-arm, prospective therapeutic trial. Pembrolizumab (MK-3475), 200 mg IV Q3W starting at C1D1/Week 1 for up to 2 years, until disease progression, or treatment intolerance. RT, 8 Gy x 3 fractions over 3 consecutive days at C1D8/Week 2; Axatilimab (SNDX-6352; INCA034176), 1 mg/kg, IV, Q2W starting 1 week post- RT C1D15/Week 3 until disease progression or treatment intolerance.

DETAILED DESCRIPTION:
Checkpoint blockade-mediated immunotherapy (IO) is an emerging cornerstone in the treatment of triple negative breast cancer (TNBC) in both the metastatic and curative intent settings. Initial studies of IO monotherapy in heavily pretreated metastatic TNBC were disappointing with low objective response rate (ORR) (5.3%: KEYNOTE-086, KEYNOTE-119) and no effect in OS (1-3). However, recent studies in patients with previously untreated metastatic TNBC, showed IO combinations with chemotherapy were associated with improved progression-free survival (PFS) and overall survival (OS) compared to chemotherapy alone in patients with "PD-L1 positive" disease (IMpassion130 and KEYNOTE-355) (4-7). Nonetheless, nearly half of patients on IMpassion130 had grade 3 or higher toxicity, leading to a discontinuation rate of 16.9%, and over 70% of all patients on first-line IO containing regimens will experience disease progression within one year. Based on these data, IO-containing regimens have become the standard-of-care treatment option for metastatic TNBC, albeit with a high failure rate and a non-trivial toxicity profile. Second line antibody-drug conjugate Sacituzumab govitecan while also improving response in metastatic TNBC still has 85% of patients fail at 1 year (ASCENT, Bardia NEJM 2021). Therefore, novel strategies that augment IO-enhanced tumor-specific responses and limit treatment-associated toxicities are critically important in TNBC. Lastly, radiotherapy (RT), commonly used in palliation of metastatic TNBC, is a potent modulator of the immune response, and can produce responses in unirradiated tumors in combination with IO (8-11).

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years at the time of consent.
* Patients with metastatic or locally recurrent TNBC who received prior immunotherapy in any setting (curative or advanced/metastatic).
* Have ≥2 measurable, non-osseous, non-hepatic recurrent or metastatic lesions. Of these lesions, at least one is indicated for radiation therapy and at least one will not be irradiated to be used to determine response. Notes on lesions: patients are still eligible if they have liver or bone lesions, so long as at least 2 measurable lesions are non-osseous, non-hepatic recurrent or metastatic per above criterion.
* Histologically or cytologically-confirmed TNBC, defined as ER <10%, PR <10%, HER2-negative by ASCO CAP guidelines. Note: HER2 0-2+ IHC is allowed (i.e., if FISH-negative, this is still considered HER2-negative).
* ECOG Performance Status ≤ 1.
* Demonstrate adequate organ function
* Female subject of childbearing potential should have a negative serum or urine pregnancy test or documentation of absence of pregnancy by a gynecologist within 14 days of initiating first dose of pembrolizumab for eligibility verification.
* Female subjects of childbearing potential should be willing to use highly effective contraceptive methods (Appendix 12.6) during the treatment period through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male participants should be willing to use highly effective contraceptive methods (Appendix 12.6) during the treatment period through 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria

* Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
* Is currently participating and receiving study therapy, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has had prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study treatment Day 1 or who has not recovered (i.e., > Grade 1 or baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy or targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., > Grade 1 or baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Has a known additional malignancy that is progressing or has required treatment within the last 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤6, and PSA <10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least four weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.).
* Has known history of/active, non-infectious pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/active interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment. Note: Negative urine or serum pregnancy test is also conducted within 72 hours prior to C1D1 for study procedures but if screening pregnancy test is done within 72 hours of C1D1, it is not required to be repeated.
* Has a known history of Human Immunodeficiency Virus (HIV). HIV testing is not required unless mandated by local health authority.
* History of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as detectable HCV RNA [qualitative]) infection. Note: Testing for Hepatitis B or C is not required unless mandated by local health authority.
* Has received a live vaccine or live-attenuated vaccine within 30 days of planned start of pembrolizumab. Administration of killed vaccines is allowed.
* Has had an allogeneic tissue/solid organ transplant, including patients with prior allogeneic hematopoietic stem-cell transplant.
* Patients eligible for PARP inhibitor therapy.
* Any patient with prior immune-related treatment toxicity for which permanent discontinuation is indicated.
* History of acute or chronic pancreatitis. Note: Participants who had a defined pancreatitis etiology (e.g., pancreatitis due to gallstones, trauma/injury, or medications such as asparaginase) may be enrolled if pancreatitis resolved prior to study enrollment.
* History of thromboembolic events (such as deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction) in the 6 months prior to study enrollment.
* Currently active significant cardiac disease, such as uncontrolled arrhythmias, uncontrolled hypertension, or Class 3 or 4 congestive heart failure as defined by New York Heart Association, or a history of myocardial infarction or unstable angina within 6 months prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From start of study treatment until subject proceeds to standard of care treatment, up to 2 years.
  The proportion of patients with confirmed PR or CR per RECIST v1.1, assessed from the start of study treatment (defined as from first dose of pembrolizumab) for up to two years. ORR in the non-targeted, unirradiated lesion(s) as defined by CR or PR per iRECIST. Objective response will be assessed separately in all sites that are not irradiated.

SECONDARY OUTCOMES:
Number of Adverse Events Related to Study Treatment | From start of study treatment up to 90 days post end of study treatment.
  To determine the safety, toxicity, and tolerability of the combination in recurrent or metastatic TNBC. Safety, toxicity, and tolerability of the combination will be assessed by the number of adverse events related to study treatment per NCI's CTCAE v5.0 from start of study treatment up to 90 days post end of study treatment.
Progression-free survival (PFS) | Up to 2 years post end of study treatment.
  To assess progression-free survival (PFS). Assessed from the start of study treatment until documented progression, or death due to any cause.
Overall Survival (OS) | Up to 2 years post end of study treatment.
  To assess overall survival (OS). Assessed from the start of study treatment until death due to any cause.
Duration of Response (DoR) | Up to 2 years post end of study treatment.
  To assess duration of response (DoR). Assessed from the start of study treatment until documented progression, or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shiao, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No